CLINICAL TRIAL: NCT02698969
Title: Recovery of Muscle Function After Deep Neuromuscular Block by Means of Dia-phragm Ultrasonography and Adductor Pollicis Acceleromyography: Comparison of Neostigmine vs. Sugammadex as Reversal Drugs.
Brief Title: Recovery of Muscle Function After Deep Neuromuscular Block by Means of Diaphragm Ultrasonography
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Chiara Adembri, Medical Doctor, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUDRACT 2013-004-787-62
Record Dates: First submitted 2016-02-15; First posted 2016-03-04 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Post-operative Residual Curarization
Keywords: Sugammadex; Post-operative residual curarization; Diaphragm Ultrasonography
MeSH Terms: interventions — Sugammadex; Neostigmine; Atropine; Rocuronium; Fentanyl; Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugammadex (Experimental): patients enrolled who will receive sugammadex 2 mg*kg-1 at the end of surgery
  Interventions: Drug: Sugammadex; Device: Diaphragm Ultrasonography; Device: Neurumuscual monitoring; Drug: Rocuronium; Drug: Fentanyl; Drug: Propofol; Drug: Sevoflurane
- Nestigmine, Atropine (Active Comparator): patients enrolled who will receive neostigmine 50 mcg*kg-1 and atropine 15 mcg*kg-1 at the end of surgery
  Interventions: Device: Diaphragm Ultrasonography; Drug: Neostigmine; Drug: Atropine; Device: Neurumuscual monitoring; Drug: Rocuronium; Drug: Fentanyl; Drug: Propofol; Drug: Sevoflurane

INTERVENTIONS:
Drug: Sugammadex
  Other Names: Bridion
  Arms: Sugammadex
Device: Diaphragm Ultrasonography — Prior to induction of anesthesia each enrolled patients, ultrasonography diaphragm evaluation will be performed using an ESAOTE ultrasound machine (ESAOTE MyLab, Genova, Italy) by assessing the TF and amplitude of excursion.
  Other Names: Diaphragm Ultrasound
Drug: Neostigmine
  Other Names: Prostigmin
  Arms: Nestigmine, Atropine
Drug: Atropine
  Arms: Nestigmine, Atropine
Device: Neurumuscual monitoring — Neuromuscular monitoring assesses muscle recovery after deep neuromuscular block through trainf of four and post tetanic count method
  Other Names: Train of Four and post tetanic count
Drug: Rocuronium — Rocuronium will be administered 0.6 mg*kg-1 to reach neuromuscular block at the induction of general anesthesia and 0.15 mg*kg-1 when PTC elicits more than 5 twitches in order to maintain a deep neuromuscular block
  Other Names: Esmeron
Drug: Fentanyl — Fentanest will be administered 2 mcg*kg-1 at the induction of general anesthesia and titrated 0.5 mcg*kg-1 every 30 minutes
  Other Names: Fentanest
Drug: Propofol — Propofol will be administered 2 mg*kg-1 at the induction of general anesthesia
  Other Names: Diprivan
Drug: Sevoflurane — Sevoflurane will be administered at 1.0 MAC in an air/oxygen mixture
  Other Names: Sevorane

SUMMARY:
Diaphragm ultrasonography as a diagnostic tool in order to demonstrate the superiority of Sugammadex vs. AChEI in facilitating post-operative neuromuscular recovery.

DETAILED DESCRIPTION:
The proposed study will be a prospective, double-blind, single center randomized study performed in 60 patients with ASA physical status I-II, between 18-80 years old, undergoing dNMB with rocuronium during ear nose and throat (ENT) surgery. Randomization will be performed using a table created from the website www.randomization.com, and patients will be divided equally into two groups: Treatment with Sugammadex (SUG group) or treatment with Neostigmine (NEO group). Exclusion criteria will include: A history of hepatic or renal disease, chron-ic or acute alcoholism, allergy or hypersensitivity to Sugammadex and/or atropine or Neostigmine, current medications with CNS effects, a history of neurologic disease, diaphragmatic palsy, pregnancy or nursing arrhythmias. Continuous neuromuscular monitoring will be performed using TOF ratios obtained from ad-ductor pollicis muscle. At the conclusion of the surgical procedure, patients will receive either Neostigmine (NEO group) or Sugammadex (SUG group) for NMB reversal. The physician who will administer the study drugs will insure that is per-formed on an open-label (non-blinded) basis. All patients showing a TOF ratio ≥0.9 will be extubated. Diaphragmatic function (assessed by ultrasonographic evaluation of the TF and amplitude of excursion) will be evaluated in each subject at the following time points:

1. Prior to induction of general anesthesia.
2. At the conclusion of the surgical procedure when TOF ratio is 0.9.
3. 15 and 30 minutes after discharge from the operating theatre. The physician who will perform the ultrasound scan will be different from the one who involved with administration of the drug for NMB reversal and the former will be blinded with respect to treatment received by patients. It is likely that, despite a TOF value greater than 0.9, higher diaphragm recovery will occur earlier and last longer when reversal of the NMB is achieved using Sugammadex (a specific antagonist) when compared with Neostigmine (a non-specific reversal).

In order to standardize the anesthetic technique, no premedication will be administered to any patient candidate to undergo to microlaryngoscopy procedure. Besides each individual enrolled will receive neuromuscular monitoring with ulnar nerve stimulation with TOF Watch® (Organon, Oss, Netherlands). The device will be calibrated pre-operatively and parameters set using standard train of four (TOF) methodology after administration of hypnotic drug prior to muscle relaxation. Standard induction of general anesthesia will be performed using intravenous (iv) fentanyl (2 mcg kg-1), propofol (2 mg kg-1), and rocuronium (0.6 mg kg-1). Tracheal intubation will be performed when the patient fails to register signals with TOF. Rocuronium (0.15 mg kg-1) will be re-administered when PTC elicits more than 5 twitches in order to maintain a dNMB. Sevoflurane will be administered at1.0 MAC in an air/oxygen mixture. Fentanyl will be titrated with a bolus of 0.5 mcg kg-1 every 30 minutes to maintain analgesia. Prior to induction of anesthesia, ultrasonography diaphragm evaluation will be performed using an ESAOTE ultrasound machine (ESAOTE MyLab, Genova, Italy) by assessing the TF and amplitude of excursion. With the spontaneously breathing patient in semi-recumbent position, the amplitude of excursion will be evaluated following the method of Kim et al (7) using a 3.5-MHz ultrasound probe placed over the intercostal space above the 10th rib in the right mid-axillary line for the right diaphragm and the left mid-axillary line for the left diaphragm. The liver or spleen will be used as a window for each hemi-diaphragm. A two-dimensional mode will be used to find the best approach and to select the exploration line of each hemi-diaphragm. With the probe fixed on the chest wall during respiration, the ultrasound beam will be directed to the hemi-diaphragmatic domes at an angle of not less than 70°. During inspiration, the normal diaphragm contracts and moves caudally toward the transducer; this will be recorded as an upward motion of the M-mode tracing. The amplitude of excursion will be measured on the vertical axis of the tracing from the baseline to the point of maximum height of inspiration on the graph. Three measurements will be performed for each patient and averaged for each side at each time point of the protocol (7). Moreover, TF will be assessed following the method of Vivier et al (6) with a linear high frequency probe set at 12 Mhz. The diaphragm will be located with same method described above and the zone of apposition will assessed at 0.5-2 cm below the costophrenic sinus. The inferior border of the costophrenic sinus will be identified at end-inspiration as the zone of transition from the artifact representation of normal lung (the lung sliding) to the visualization of diaphragm and liver.

The diaphragm thickness will be recorded in time motion (TM) mode. The diaphragm will be outlined using the two clear bright parallel lines of the pleural and peritoneal membranes. Measurements will be averaged out of three or more consecutive breaths on the last valid image recorded at the end of each period (6) .At the conclusion of the surgical procedure and when TOF neuromuscular monitoring shows a minimum of 2 twitches, patients will randomly receive, as described above, either (NEO Group) iv Neostigmine 50 µg kg-1 and atropine 15 µg kg-1 or (SUG group) iv Sugammadex 2 mg kg-1 to reverse residual curarization. Extubation will be performed when all of the following criteria are met: Patient is awake and executes simple commands, shows regular respiratory pattern with a tidal volume of 6-7 mL/kg referred to ideal body weight (IBW) and a TOF ratio ≥0.9. During the period preceding a TOF ratio > 0.9 , bilateral diaphragm ultrasonography evaluating amplitude of excursion and TF will be performed to assess muscle recovery in spontaneous breathing patients. These measurements will be compared with baseline muscle assessment. Three additional diaphragm ultrasound scans will be performed 15 and 30 minutes after discharge from operating theatre. Follow up will be performed to document every adverse event and complication that occurs until discharge from the hospital.

Data will be collected by the use of paper CRF pages. Data entry will be performed at one central site that will maintain the overall database and will perform and be responsible for the data analysis.

The study will be conducted within 8 months -1 year from approval from our ethical committee. A preliminary report will be completed and submitted after the first six months of data collection.

Data will be collected by the use of paper CRF pages. Data entry will be performed at one central site that will maintain the overall database and will perform and be responsible for the data analysis. All the compiled CRFs will be archived. In order to eliminate possible data entry errors, individual data will be compared to a range of plausible values. After data entry, automated checks, that are defined beforehand (a priori), will be performed to evaluate internal inconsistencies, range errors, or missing data. For each atypical/out-of-range/missing data, a query will be automatically sent to the investigator. Once all the queries are solved, the database will be locked and used for statistical analysis.Statistical analysis will be performed in collaboration by the Department of Statistics of the University of Florence. Complete data will not be unblinded until the external medical and statistics review have been completed.

Data will be collected and a single statistical analysis will be performed at the completion of the study using an intention to treat (ITT) analysis. With regard to the primary endpoint, differences between the two groups with respect to distribution of muscle function recovery after deep muscular blockade will be subjected to non-parametric tests depending on the characteristics of outcome distribution. To compare the primary endpoint between the 2 groups, the data will be analysed using Wilcoxon rank sum test for two independent samples as they are expected to be continuous and not normally distributed. As a sensitivity analysis, parametric tests will potentially be employed after thorough evaluation of the validity distribution assumptions.

The ultrasonography and TOF data will be summarized by drug treatment group as mean, standard deviation, quintiles, and minim and maximum values. In addition, two-sided 95% confidence intervals will be calculated on the comparison between the two groups for the main descriptive parameters of the primary and secondary variables.

In order to compare the different percentage of respiratory events in the two arms studied, a chi square test will be performed.

Finally, descriptive statistics of all variables describing characteristics of the patients enrolled in the study and of patients excluded from the study will be produced. The mean, median, standard deviation and range will be calculated for continuous data by drug treatment group. For categorical variables, frequency counts and percentages will be calculated.

Power/Sample Size:

Because this is the first clinical trial that proposes to evaluate this endpoint, no published data are available at this time. However, assuming a 25% of difference of TF between groups would be clinically meaningful, a confidence interval of 95% and power 80%, sample size calculation provided by StatCalc EPI INFO ver 7.0 (Center for Diseases Control, Atlanta, GA, USA) considered 28 patients for each group fundamental to reach the endpoint predefined. This proposal requests funding for a pilot study, with a double blind design, where participants will be randomly enrolled to receive Sugammadex or Neostigmine with a 1:1 allocation using the standardized table created with the website www.randomization.com.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* age between 18-80 years old
* dNMB with rocuronium during ear nose and throat (ENT) surgery

Exclusion Criteria:

* Clinical diagnosis of hepatic or renal disease
* Clinical diagnosis of chronic or acute alcoholism
* History of allergy or hypersensitivity to Sugammadex and/or atropine or Neostigmine
* Current medications with CNS effects
* History of neurologic disease
* Diaphragmatic palsy
* Pregnancy or nursing
* History of malignant arrhythmias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-operative residual curarization (PORC) as assessed by diaphragm ultrasonography in order to determine its muscle strenght | 30 minutes from the end of surgical procedure
  The clinician will assess TF (defined as a percentage) and amplitude of excursion (expressed in millimetres) of the diaphragm by means of ultrasonography

SECONDARY OUTCOMES:
Number of participants with post-operative complications related to PORC such as pneumonia as assessed chest x ray, drop of SpO2 by means of pulse oximeter and blood gas sample. | up to 1 week
Number of participants with post-operative nausea and vomiting (PONV) as assessed by postoperative nause and vomiting visual analogic scale (PONV VAS) | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Adembri, MD, Principal Investigator — University of Florence
Locations (1):
- Azienda Ospdaliero Universitaria Careggi, Florence, Italy

REFERENCES:
- [Result] Viby-Mogensen J. Postoperative residual curarization and evidence-based anaesthesia. Br J Anaesth. 2000 Mar;84(3):301-3. doi: 10.1093/oxfordjournals.bja.a013428. No abstract available. PMID 10793585
- [Result] Naguib M, Kopman AF, Ensor JE. Neuromuscular monitoring and postoperative residual curarisation: a meta-analysis. Br J Anaesth. 2007 Mar;98(3):302-16. doi: 10.1093/bja/ael386. PMID 17307778
- [Result] Flockton EA, Mastronardi P, Hunter JM, Gomar C, Mirakhur RK, Aguilera L, Giunta FG, Meistelman C, Prins ME. Reversal of rocuronium-induced neuromuscular block with sugammadex is faster than reversal of cisatracurium-induced block with neostigmine. Br J Anaesth. 2008 May;100(5):622-30. doi: 10.1093/bja/aen037. Epub 2008 Apr 2. PMID 18385265
- [Result] Wait JL, Nahormek PA, Yost WT, Rochester DP. Diaphragmatic thickness-lung volume relationship in vivo. J Appl Physiol (1985). 1989 Oct;67(4):1560-8. doi: 10.1152/jappl.1989.67.4.1560. PMID 2676955
- [Result] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Derived] Cappellini I, Ostento D, Loriga B, Tofani L, De Gaudio AR, Adembri C. Comparison of neostigmine vs. sugammadex for recovery of muscle function after neuromuscular block by means of diaphragm ultrasonography in microlaryngeal surgery: A randomised controlled trial. Eur J Anaesthesiol. 2020 Jan;37(1):44-51. doi: 10.1097/EJA.0000000000001055. PMID 31356374
- [Derived] Cappellini I, Picciafuochi F, Ostento D, Danti G, De Gaudio AR, Adembri C. Recovery of muscle function after deep neuromuscular block by means of diaphragm ultrasonography and adductor of pollicis acceleromyography with comparison of neostigmine vs. sugammadex as reversal drugs: study protocol for a randomized controlled trial. Trials. 2018 Feb 21;19(1):135. doi: 10.1186/s13063-018-2525-7. PMID 29467022